CLINICAL TRIAL: NCT00701727
Title: Ezetimibe Reverse Cholesterol Transport (RCT) Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radiant Research (Other)
Responsible Party: Michael H. Davidson, MD, FACC, Radiant Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Ezetimibe RCT-001
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-03

CONDITIONS: Hypercholesterolemia
Keywords: metabolic diseases; metabolic disorder; dyslipidemias; lipid metabolism disorders
MeSH Terms: conditions — Hypercholesterolemia; Metabolic Diseases; Dyslipidemias; Lipid Metabolism Disorders | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ezetimibe (10mg/day)for 7 weeks
  Interventions: Drug: ezetimibe
- 2 (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ezetimibe — 1 tablet,10mg, once a day, for 7 weeks
  Arms: 1
Drug: Placebo — 1 tablet, once a day, for 7 weeks
  Arms: 2

SUMMARY:
This is a prospective, placebo-controlled, cross-over trial comparing the the effects of approximately 7 weeks of placebo treatment to 7 weeks of ezetimibe (10mg/day) treatment on several parameters of reverse cholesterol transport (RCT) in men and post-menopausal women diagnosed with hypercholesterolemia. The primary hypothesis is that the ezetimibe treatment will increase the excretion of endogenous (plasma-derived) cholesterol as fecal sterols, with secondary hypotheses that there will be a significant increase in de novo cholesterol synthesis, treatment will increase cholesterol efflux from tissues into the bloodstream, and increase global RCT.

DETAILED DESCRIPTION:
The study will compare the effects of approximately 7 weeks of placebo treatment to 7 weeks of ezetimibe (10mg/day) on: 1) the efficiency of endogenous (plasma-derived) cholesterol excretion (%/day) 2) de novo cholesterol (DNC) synthesis ((%/day) 3) cholesterol efflux from tissues into blood (Ra), and 4) global RCT (efflux from tissues that is excreted as fecal sterols). Subjects will receive 7 weeks of either treatment or placebo, undergo RCT and DNC measurements, taking 10 days, then cross-over to the alternate placebo or treatment for an additional 7 weeks, followed by a second set of RCT and DNC measurements.

ELIGIBILITY:
Inclusion Criteria:

* male, non-smoker, 21-75 years of age
* female, non-smoker, 40-75 years of age
* post-menopausal women, as defined by lack of menses for at least 2 years and age >55, OR history of documented bilateral oophorectomy, confirmed with an elevated FSH at screening
* low-density lipoprotein (LDL) concentration between 130-200 mg/dL.
* triglyceride (TG) concentration <350 mg/dL, inclusive
* high-density lipoprotein (HDL) between 30-60 mg/dL for men and 40 -70 mg/dL for women
* ability to give informed consent

Exclusion Criteria:

* Subject has history of diabetes mellitus, active hepatitis, gall bladder disease, gastric or ileal bypass surgery, irritable bowel syndrome, and gastrointestinal disorder/condition associated with malabsorption, or clinically significant abnormalities on screening (prestudy) physical examination of laboratory tests.
* Screening laboratory tests with hematocrit <30%, aspartate aminotransferase/alanine aminotransferase (AST/ALT) >2*upper limit of normal, abnormal thyroid-stimulating hormone (TSH), fasting glucose >=126mg/dL
* renal impairment with creatinine clearance (CRCl)<80ml/min
* treatment within the last 2 months with drugs known to alter lipid metabolism including beta blockers, thiazide diuretics, bile acid resins, statins, ezetimibe, niacin, fibrates, plant stanol esters (eg Benecol,phyto sterols) and fishoils
* history of known coronary heart disease (CHD), stroke or prior revascularization procedure or peripheral vascular disease
* history of allergy to egg or soy products
* current or recent (past 12 months) of drug abuse or alcohol abuse. Alcohol use must be limited to no more than 2 drinks/day (1 drink=12 oz beer, 5 oz wine, or 1.5 oz hard liquor). Subject must be willing to avoid large day-to-day fluctuations in alcohol intake.
* participation in another clinical trial or exposure to any investigational agent within 30 days prior to Visit 1
* Individual has a condition the Principal Investigator believes would interfere with his/her ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results, or put the subject at undue risk

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Davidson, Md. FACC, Principal Investigator — Radiant Research
Locations (1):
- Radiant Research, Chicago, Illinois, United States

REFERENCES:
- [Derived] Davidson MH, Voogt J, Luchoomun J, Decaris J, Killion S, Boban D, Glass A, Mohammad H, Lu Y, Villegas D, Neese R, Hellerstein M, Neff D, Musliner T, Tomassini JE, Turner S. Inhibition of intestinal cholesterol absorption with ezetimibe increases components of reverse cholesterol transport in humans. Atherosclerosis. 2013 Oct;230(2):322-9. doi: 10.1016/j.atherosclerosis.2013.08.006. Epub 2013 Aug 13. PMID 24075764

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited at a research clinic, Chicago, IL, from June 2008 to October 2008
Pre-assignment Details: 61 subjects screened, 30 subjects excluded(8 failed inclusion criteria, 9 failed exclusion criteria, 3 had unsuitable veins, 5 failed a drug screen, 1 was lost-to-follow-up, 4 were excluded when enrollment was complete), 31 subjects randomized.
Groups:
- Ezetimibe First, Placebo Second: Ezetimibe first for 7 weeks, followed by placebo for 7 weeks
- Placebo First, Ezetimibe Second: Placebo first for 7 weeks,followed by ezetimibe for 7 weeks
Period: First Treatment Period
Arm/Group | Ezetimibe First, Placebo Second | Placebo First, Ezetimibe Second
Started | 16 | 15
Completed | 15 | 13
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — sponsor decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Second Treatment Period
Arm/Group | Ezetimibe First, Placebo Second | Placebo First, Ezetimibe Second
Started | 15 | 13
Completed | 13 | 13
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive ezetimibe first and placebo first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Fecal Excretion of Plasma-derived Cholesterol
Description: (Fecal excretion of plasma-derived cholesterol):The following measurements will be made following isotope infusion:
  1. The composition of fecal neutral and acidic sterols will be measured as % of total.
  2. The excretion rate of fecal neutral and acidic sterols will be measured as mg/day.
  3. The isotopic enrichment of both fecal neutral and acidic sterols will be measured as atomic percent excess (% APE).
  4. Fecal isotope excretion, or recovery, of plasma-derived cholesterol will be calculated as %/day.
Time Frame: 7 weeks
Population: Per Protocol,all subjects
Measure: Mean (Standard Deviation); unit: mg/day cholesterol excreted
Groups:
- Placebo: placebo daily,7 weeks
- Ezetimibe: Ezetimibe 10 mg/day 7 weeks
Arm/Group | Placebo | Ezetimibe
Number analyzed (Participants) | 26 | 26
mg/day cholesterol excreted | 1593 (1287) | 1950 (915)
Statistical Analysis 1: Comparison: Placebo vs Ezetimibe; Test type: Superiority or Other; p = 0.019, t-test, 2 sided

2. Secondary Outcome: Change From Baseline in Total Cholesterol, From Fasting Plasma Samples
Description: plasma levels of total cholesterol
Time Frame: 7 weeks
Population: per protocol, all subjects
Measure: Mean (Standard Deviation); unit: mg/dL total cholesterol
Arm/Group | Placebo | Ezetimibe
Number analyzed (Participants) | 26 | 26
mg/dL total cholesterol | 219 (26) | 187 (24)
Statistical Analysis 1: Comparison: Placebo vs Ezetimibe; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: de Novo Cholesterol Synthesis (DNC)
Description: Plasma DNC will be measured following the isotope infusion of deuterated water, expressed as %.
Time Frame: 7 weeks
Population: per protocol, all subjects
Measure: Mean (Standard Deviation); unit: %/day plasma DNC
Arm/Group | Placebo | Ezetimibe
Number analyzed (Participants) | 26 | 26
%/day plasma DNC | 3.4 (0.1) | 4.7 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Ezetimibe; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Cholesterol Efflux Rate (Ra Cholesterol)
Description: The efflux, or mobilization, rate of cholesterol from peripheral tissues into the plasma will be measured as mg/kg/hr. An IV infusion of [13C2] cholesterol mixed in 10% Intralipid® and 10 % ethanol is given piggy-backed into normal saline over 20 hours (4pm - 12 noon). This is used to determine rate of appearance (Ra) cholesterol, which will be measured by dilution of infused [13C2] cholesterol during the plateau phase of plasma enrichment (approximately the last 4 hours of the infusion), as well as to provide the plasma cholesterol that will be traced into biliary sterols.
Time Frame: 7 weeks
Population: per protocol, all subjects
Measure: Mean (Standard Deviation); unit: mg/kg/hr cholesterol
Arm/Group | Placebo | Ezetimibe
Number analyzed (Participants) | 26 | 26
mg/kg/hr cholesterol | 4.6 (0.5) | 4.4 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Ezetimibe; Test type: Superiority or Other; p = 0.12, t-test, 2 sided

5. Secondary Outcome: Triglycerides (TG)
Description: Change from baseline in plasma triglycerides, measured in fasting blood samples
Time Frame: 7 weeks
Population: per protocol, all subjects
Measure: Mean (Standard Deviation); unit: mg/dL TG
Arm/Group | Placebo | Ezetimibe
Number analyzed (Participants) | 26 | 26
mg/dL TG | 128 (48) | 121 (50)
Statistical Analysis 1: Comparison: Placebo vs Ezetimibe; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

6. Secondary Outcome: Low-density Lipoprotein (LDL);
Description: Change from baseline in plasma low-density lipoprotein(LDL), measured in fasting blood samples
Time Frame: 7 weeks
Population: per protocol, all subjects
Measure: Mean (Standard Deviation); unit: mg/dL LDL
Arm/Group | Placebo | Ezetimibe
Number analyzed (Participants) | 26 | 26
mg/dL LDL | 148 (24) | 116 (20)
Statistical Analysis 1: Comparison: Placebo vs Ezetimibe; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

7. Secondary Outcome: High-density Lipoprotein (HDL)
Description: Change from baseline in plasma HDL, measured in fasting blood samples
Time Frame: 7 weeks
Population: per protocol, all subjects
Measure: Mean (Standard Deviation); unit: mg/dL HDL
Arm/Group | Placebo | Ezetimibe
Number analyzed (Participants) | 26 | 26
mg/dL HDL | 46 (9) | 45 (11)
Statistical Analysis 1: Comparison: Placebo vs Ezetimibe; Test type: Superiority or Other; p = 0.95, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 7 weeks
Groups:
- Placebo: Placebo, 10 mg/day, for 7 weeks
- Ezetimibe: ezetimibe, 10 mg/day, for 7 weeks
Arm/Group | Placebo | Ezetimibe
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 15/31 | 15/31
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | Ezetimibe (N=31)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No